CLINICAL TRIAL: NCT05811858
Title: Analyzing Factors Impacting Patient Involvement in Osteoarthritis Clinical Research
Brief Title: Investigating Medical Research Trends in Osteoarthritis Clinical Trials
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 84129695
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical research participation percentages haven't always been fully representative of a given demographic.

The goal is to find out which aspects of a clinical trial may make it more difficult for patients to take part or see it through.

The data will be evaluated through different demographic lenses and identify trends that could help improve the experience of future osteoarthritis patients during clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed.
* Participant has a diagnosis of osteoarthritis.
* Willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.

Exclusion Criteria:

* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent.
* Pregnant or lactating woman
* Known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug(s) administration or interfere with the interpretation of safety results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with osteoarthritis who are actively considering involvement in an observational clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in an osteoarthritis clinical study. | 3 months
Number of osteoarthritis patients who remain in clinical trial until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stabile M, Van Ryssen B, Minei S, Coppieters E, Crovace A, Lacitignola L, Staffieri F. Observational study of the clinical value of the canine osteoarthritis staging tool. Vet J. 2022 May-Jun;283-284:105832. doi: 10.1016/j.tvjl.2022.105832. Epub 2022 Apr 27. PMID 35487477
- [Background] Akesson KS, Sunden A, Stigmar K, Fagerstrom C, Pawlikowska T, Ekvall Hansson E. Enablement and empowerment among patients participating in a supported osteoarthritis self-management programme - a prospective observational study. BMC Musculoskelet Disord. 2022 Jun 8;23(1):555. doi: 10.1186/s12891-022-05457-9. PMID 35676666
- [Background] Ellis KR, Cuthbertson CC, Carthron D, Rimmler S, Gottfredson NC, Bahorski SG, Phillips A, Corbie-Smith G, Callahan L, Rini C. A Longitudinal Observational Study of Multimorbidity and Partner Support for Physical Activity Among People with Osteoarthritis. Int J Behav Med. 2021 Dec;28(6):746-758. doi: 10.1007/s12529-021-09985-x. Epub 2021 Apr 2. PMID 33797056

DOCUMENTS (1):
  • Informed Consent Form (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT05811858/ICF_000.pdf